CLINICAL TRIAL: NCT05884892
Title: Egyptian Hypertrophic Cardiomyopathy Program
Status: Recruiting | Type: Observational
Sponsor: Magdi Yacoub Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AHC-HCM
Record Dates: First submitted 2022-12-14; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: HCM; HOCM; Hypertrophic Cardiomyopathy; Familial Hypertrophic Cardiomyopathy; Hypertrophic Cardiomyopathy with Genetic Marker; Hypertrophic Obstructive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathy, Hypertrophic, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Our biobank includes:
  * Blood samples for genetic analysis from all recruited patients and their family members.
  * Human specimens collected from hypertrophic cardiomyopathy patients after surgical intervention (extended septal myectomy).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Egyptian HCM program aims at defining incidence, severity, phenotype, genotype and determinants of the disease in Egypt, and providing state-of-the-art treatment strategies including medical, surgical and interventional procedures which are patient- and disease-specific.

DETAILED DESCRIPTION:
This project aims to:

* Define incidence, severity, phenotype, genotype and determinants of the disease in Egypt.
* Characterise the phenotype and genotype of several large cohorts with inherited muscle disease and their relatives.
* Provide state-of-the-art treatment strategies including medical, surgical and interventional procedures which are patient- and disease-specific.
* Study the basic mechanisms responsible for the different phenotypes at a molecular and cellular level including genotype-phenotype correlation.
* Provide a special focus for studying patients who are genotype positive and phenotype negative which we believe could yield critical data regarding the evolution of the disease.
* Develop sophisticated laboratory studies for single cell electrophysiology and immunocytochemistry and others focusing on the explanted human material from the surgical program.
* Define the role of microvascular coronary artery in the development and progression of the disease.
* Training Egyptian cardiologists, cardiac surgeons and scientists on state-of-the-art diagnosis and management of heart muscle disease including the latest developments in imaging, novel surgical techniques, coronary physiology, next generation sequencing, bioinformatics and cellular electrophysiology.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with hypertrophic cardiomyopathy (index patients) who are willing and consented to participate in the registry.
* All family members of index patients who are willing and consented to participate in the registry.

Exclusion Criteria:

* Refusal to consent to participate in the registry program.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian patients diagnosed with hypertrophic cardiomyopathy (either obstructive or non-obstructive), and their family members (either apparently healthy or not) who are willing to participate in this registry.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of HCM in Egypt | through study completion, an average of 5 year
  per 100,000 population per year
Determinants of clinical severity of HCM in Egypt | through study completion, an average of 1 follow-up every year, and an average of 5 follow-ups throughout the study duration
  Several indicators describing the clinical symptoms and signs
Determinants of cardiac phenotype severity of HCM in Egypt | through study completion, an average of 1 follow-up every year, and an average of 5 follow-ups throughout the study duration
  Several indicators describing the cardiac phenotype using multimodality imaging
Determinant of genotype severity of HCM in Egypt | through study completion, at least once at the time of inclusion
  To identify and report the genetic profile of HCM in Egypt.
Study the basic mechanisms responsible for the HCM in Egypt | through study completion, at least once at the time of inclusion, or
  To study different phenotypes at a molecular and cellular level including genotype-phenotype correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan Heart Centre - Magdi Yacoub Heart Foundation, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided